CLINICAL TRIAL: NCT04451824
Title: Contour Research CL-100 Examination of Circumferential Reduction: A Review of Data Collected From Routine Use of the Device
Brief Title: Examination of Circumferential Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contour Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL100 CR RetrX1
Record Dates: First submitted 2020-06-16; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Routine use of device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention with Routine Use of Red Light (Experimental): Routine Use of red light (635nm) for 30 minutes on patients is to be observed in relation to its effect(s) in achieving circumferential reduction of the thighs, hips and waist of the patient, and a contour reduction of any protrusion of fat.
  Interventions: Device: CL-100

INTERVENTIONS:
Device: CL-100 — Red Light LED device for circumferential reduction

SUMMARY:
The rationale for the selection of Outcome Measures is the compliance with FDA regulations as pertain to medical devices with a moderate level of risk of hazard leading to harm of the patient; firstly, the safety of the device in achieving the desired effect of its intended use when operated in the intended manner; and secondly, the effectiveness of the device in achieving its desired effect of its intended use in accordance with its proposed label and labeling. The rationale for the selection of the primary outcome measure is to satisfy the question of safety and effectiveness of the use of red-light exposure to reduce the circumference of overweight patients with a statistically significant Routine Use population size. Given that the Routine Use Data Analysis is open label and therefore not blinded, there is no need for a control group nor additional cohorts for varying levels of exposure and corresponding safety and/or effectiveness.

DETAILED DESCRIPTION:
In the 1960s, the concept of using light energy for a variety of health maintenance goals and overcoming a number of dermatological conditions began in earnest to receive the attention of NASA researchers as a means of providing desired clinical outcomes to astronauts while in the confines of a space capsule over long periods of time. The research was well funded and supported by the U.S. government, and confirmed the value of light emitting diode (LED) low-level light therapy (LLLT), in particular red light from the 635nm frequency, for producing a variety of healthful effects within the dermis. The ability to achieve a reduction in the dimensions of exposed liposomes using red light is intended to be confirmed by analyzing the clinical data from a minimum of one hundred patients who were exposed to the 635 nm frequency for 30 minutes by use of the subject device (Contour Light) during routine use to confirm that the device is safe and effective for its intended application. Please see the following clinical articles, appended in section 10.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females ages 18 and above
* Generally good health

Exclusion Criteria:

* Pregnancy
* Active cancer within the past year
* Pacemaker
* Diminished ability to void waste (liver and/or kidney function impairment)
* Photosensitivity (generally and/or from medication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Examination of Circumferential Reduction - Primary Objective | <1 hour
  To confirm the proper use of the device induces a change in the circumference of the patients thighs, hips and waist, when exposed to the red light (635nm)

SECONDARY OUTCOMES:
Examination of Circumferential Reduction - Secondary Objective | <1 hour
  To achieve a contour change, specifically a lessening of the protrusion of body fat, when exposed to the red light (635nm)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Dreier, BS, Principal Investigator — Contour Research, LLC
Locations (3):
- United States (3):
  - Gibson Clinic, Vista, California
  - Barone Clinic, Savannah, Georgia
  - Love Clinic, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data with other researchers.